CLINICAL TRIAL: NCT04889820
Title: Oncologic oUTcomes of Neoadjuvant Chemotherapy for obSTructive Colon cAncer After steNt Decompression (OUTSTAND Trial); Multicenter Randomized Controlled Trial
Brief Title: Outcome of Neoadjuvant Chemotherapy for Obstructive Colon Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Kye Bong-Hyeon, Associate professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XC21MIDI0004
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Colon Cancer, Obstruction
MeSH Terms: conditions — Colonic Neoplasms; Bites and Stings | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: 1. The Control group
     * The patients who are assigned into control group take a curative surgery within 2 weeks after successful SEMS placement. And then, after recovery period, adjuvant FOLFOX chemotherapy will be administered into them. Adjuvnat FOLFOX chemotherapy will be administered every 2week during 6 months (total 12 cycles).
  2. The Experimental group
     * The patients who are assigned into the experimental group take a neoadjuvant FOLFOX chemotherapy within 2 weeks after successful SEMS placement. After three cycles of FOLFOX, they will take a curative surgery. And then, after recovery period, adjuvant FOLFOX chemotherapy will be administered into them. Adjuvnat FOLFOX chemotherapy will be administered every 2week during about 4 months (total 9 cycles). The perioperative FOLFOX chemotherapy in the experimetal group will be totally 12 cycles during 6months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Control group (Active Comparator): - The patients who are assigned into control group take a curative surgery within 2 weeks after successful SEMS placement. And then, after recovery period, adjuvant FOLFOX chemotherapy will be administered into them. Adjuvnat FOLFOX chemotherapy will be administered every 2week during 6 months (total 12 cycles).
  Interventions: Drug: Adjuvant chemotherapy; Procedure: Curative resection
- The Experimental group (Experimental): - The patients who are assigned into the experimental group take a neoadjuvant FOLFOX chemotherapy within 2 weeks after successful SEMS placement. After three cycles of FOLFOX, they will take a curative surgery. And then, after recovery period, adjuvant FOLFOX chemotherapy will be administered into them. Adjuvnat FOLFOX chemotherapy will be administered every 2week during about 4 months (total 9 cycles). The perioperative FOLFOX chemotherapy in the experimetal group will be totally 12 cycles during 6months.
  Interventions: Drug: Neoadjuvant chemotherapy; Drug: Adjuvant chemotherapy; Procedure: Curative resection

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — In this study, patients with obstructive colon cancer will be divided into two groups; in the control group, curative surgery will be performed within 2 weeks after successful SEMS placement, and in the experimental group, 3 cycles of neoadjuvant chemotherapy will be administered into patients who undergo successful SEMS placement and then curative surgery will be performed after neoadjuvnat chemotherapy. After the surgery, adjuvant chemotherapy will be administered, and total perioperative chemotherapy will be administered with 12 cycles.
  Other Names: Curative surgery
  Arms: The Experimental group
Drug: Adjuvant chemotherapy — After the surgery, adjuvant chemotherapy will be administered, and total perioperative chemotherapy will be administered with 12 cycles.
  Other Names: curative surgery
Procedure: Curative resection — After successful SEMS placement, curate resection will be performed for all enrolled patients regardless of neoadjuvant chemotherapy.

SUMMARY:
In this study, patients with obstructive colon cancer will be divided into two groups; in the control group, curative surgery will be performed within 2 weeks after successful SEMS placement, and in the experimental group, 3 cycles of neoadjuvant chemotherapy will be administered into patients who undergo successful SEMS placement and then curative surgery will be performed after neoadjuvnat chemotherapy. After the surgery, adjuvant chemotherapy will be administered, and total perioperative chemotherapy will be administered with 12 cycles. The primary end points is overall survival, also the short-term perioperative outcomes and long-term oncological outcomes will be compared between the control and experimental group. Random allocation will be carried out with the consent of patients and their guardians after successful SEMS placement, and 204 patients will be distributed between the two groups by 1:1.

DETAILED DESCRIPTION:
It is known that approximately 30-40% of colorectal cancer require emergency surgery. Of these, the colonic obstruction accounts for 80% of situations requiring emergency treatment and colon perforation appears in 20%. In patients with colorectal cancer patients who require emergency surgery, there are higher postoperative complication rates, mortality rates, and ostomy formation rate than those who do not. In aspect of oncologic outcomes, long-term survival also appears to be worse in patients undergoing emergency surgery. Despite recent active screening for colorectal cancer, some studies have reported that the proportion of colorectal cancer obstruction and perforation requiring emergency surgery still occur as before. However, research on treatments to reduce postoperative complications and to increase long-term survival for patients with symptomatic colorectal cancer requiring emergency surgery remains inadequate.

Emergency surgery cannot be avoided when colorectal perforation occurs due to colorectal cancer. Obstructive colorectal cancer has also traditionally been performed in emergency surgery with colorectal resection and ostomy composition. However, with the development of endoscopic equipment and technology, endoscopic stent (self-expandable metallic stent, SEMS) insertion has been feasible for patients with obstructive colon cancer and many researches about a bridge to surgery which means a surgery after adequate decompression and bowel lavage using SEMS placement have been reported that a bridge to surgery can reduce postoperative complications, stoma formation, and postoperative mortality in selective cases. Currently, such studies recommend the use of SEMS to improve short-term postoperative outcomes. However in aspect of long-term oncological outcomes, the results have not yet been established.

In this study, patients with obstructive colon cancer will be divided into two groups; in the control group, curative surgery will be performed within 2 weeks after successful SEMS placement, and in the experimental group, 3 cycles of neoadjuvant chemotherapy will be administered into patients who undergo successful SEMS placement and then curative surgery will be performed after neoadjuvnat chemotherapy. After the surgery, adjuvant chemotherapy will be administered, and total perioperative chemotherapy will be administered with 12 cycles. The primary end points is overall survival, also the short-term perioperative outcomes and long-term oncological outcomes will be compared between the control and experimental group. Random allocation will be carried out with the consent of patients and their guardians after successful SEMS placement, and 204 patients will be distributed between the two groups by 1:1. Through this study, we would like to identify that neoadjuvant chemotherapy followed by curative resection after successful SEMS placement for obstructive colon cancer can bring the improvement of short-term perioperative outcome and long-term oncological outcome.

ELIGIBILITY:
Inclusion Criteria:

* i. Age : 20 years old or more and lesser than 75 years old ii. Agreement of this study iii. Clinical stage II or III colon cancer with colonic obstruction which is confirmed by pathologic review and imaging study.

iv. Colon cancer located beween distal T colon and Rectosigmoid junction colon which is defined as a tumor above 15cm from anal verge.

v. Colonocopic fiding: tumor involving whole circumference of the lumen, impossible to pass endoscope through the tumor vi. SEMS placement vii. no colonic injury and successful decompression of the colon with in 48 hours after SEMS placement.

viii. ECOG performance 0-2 ix. ASA ≤ 3 x. Appropriate function of the vital organ (acceptable liver enzyme and BUN/Cr) xi. Appropriate function of hematopoietic system (platelet ≥100,000ul, neutrophil ≥2,000ul) xii. If the patient is female in fertile period, urine hCG test is negative and she has no plan of pregnancy with 6 months after the termiation of whole treatment.

xiii. If the patient is male in fertile period, he agrees with contraception during treatment period and 6 months after the termination of whole treatment.

Exclusion Criteria:

* i. any suspicious distant metastasis ii. any other primary malignant lesion iii. Clinical stage T1or T2 and N0 iv. the sign of perforation or severe ischemia requiring ememgency operation v. the complication related to SEMS placement (severe bleeding and perforation after SEMS placement) vi. ASA 4 or more vii. ECOG 3 or more viii. colonic obstruction by benign stricture ix. pregnant woman or woman who is breastfeeding x. the paitents who already enrolled into other study or are taking medicine related to any clinical trial xi. the patients who are taking sorivudine xii. the patients who are taking Tegafur/gimeracil/oteracil xiii. the patietns who have a medical history of hypersensitivity reaction to 5-FU, oxaliplatin, leucovorin,or any medication including platinum.

xiv. Inappropriate function of vital organ (impaired renal function, elevated liver enzyme, and so on ) xv. Inappropriate function of hematopoietic system (platelet <100,000ul, neutrophil < 2,000ul) xvi. Genetic problem such as galactose intolerance, Lapp lactase deficiency, or glucose-galatose malabsorption)

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | 3 years after surgery
  3-year overall survival after curative surgery

SECONDARY OUTCOMES:
postoperative complication rate | within 30 days after surgery
  postoperative ileus, reoperation rate, wound infection, ..
stoma formation rate | within 30 days after surgery
  stoma formation rate withing 30 days after surgery
pathologic result | within 30 days after surgery
  TNM stage, lymphovascular invasion, silent perforation....
recurrence rate | 3 years after surgery
  recurrent rate after curative surgery within postoperative 3 years
disease-free survival | 3 years after surgery
  disease-free survival after curative surgery within postoperative 3 years
circulating tumor DNA | 1year after surgery
  to analyze the serial patterns of ctDNA in each step of treatments including stent placement, neoadjuvant therapy, surgery, and adjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Hyeon Kye, MD.PhD., Principal Investigator — The Catholic University of Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kye BH, Kim JH, Kim HJ, Lee YS, Lee IK, Kang WK, Cho HM, Ahn CH, Oh ST. The optimal time interval between the placement of self-expandable metallic stent and elective surgery in patients with obstructive colon cancer. Sci Rep. 2020 Jun 11;10(1):9502. doi: 10.1038/s41598-020-66508-6. PMID 32528099
- [Derived] Kye BH, Kim JH, Kim HJ, Lee YS, Lee IK, Kang WK, Cho HM, Park JK, Ahn CH, Lee JI, Oh ST, Choi BJ. Oncologic oUTcomes of neoadjuvant chemotherapy for obSTructive colon cAncer after steNt decompression (OUTSTAND trial); A study protocol of multicenter non-inferiority randomized controlled trial. BMC Cancer. 2025 Feb 3;25(1):194. doi: 10.1186/s12885-025-13588-0. PMID 39901122